CLINICAL TRIAL: NCT02250794
Title: Metformin and Sitagliptin Therapy for Adult Patients With Type 2 Diabetes Admitted to the General Medical Unit
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No subjects enrolled.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14042807
Record Dates: First submitted 2014-09-18; First posted 2014-09-26 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes mellitus; inpatient management; metformin; sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination; Metformin; Insulin Glargine; Insulin Lispro; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin glargine and insulin lispro (Active Comparator): insulin glargine 0.3 units per kg and insulin lispro 0.1 units per kg with each meal
  Interventions: Drug: insulin glargine and insulin lispro
- metformin and sitagliptin (Experimental): metformin 750 mg PO twice daily and sitagliptin 100 mg PO once daily
  Interventions: Drug: metformin and sitagliptin

INTERVENTIONS:
Drug: metformin and sitagliptin — metformin 750 mg PO twice daily
  Other Names: glucophage
  Arms: metformin and sitagliptin
Drug: insulin glargine and insulin lispro — insulin glargine given once daily
  Other Names: lantus insulin
  Arms: insulin glargine and insulin lispro
Drug: metformin and sitagliptin — sitagliptin 100 mg PO once daily
  Other Names: Januvia
  Arms: metformin and sitagliptin
Drug: insulin glargine and insulin lispro — insulin lispro given three times daily with meals
  Other Names: humalog insulin
  Arms: insulin glargine and insulin lispro

SUMMARY:
The purpose of this study is to test whether a combination of two pills commonly used to treat outpatient diabetes called metformin and sitagliptin (januvia) could provide successful control of blood sugar levels in patients with type 2 diabetes during hospitalization for the treatment of a general medical condition. Both metformin and sitagliptin are currently approved by the Food and Drug Administration for the treatment of type 2 diabetes, but little experience exists for their use in hospitalized patients. The current standard practice is to use insulin injections to control blood sugar in hospitalized patients with type 2 diabetes. This study will compare the use of metformin tablets twice per day along with sitagliptin tablets once per day with daily insulin injections in patients with type 2 diabetes during hospitalization, and will study how well the blood sugar levels are controlled.

DETAILED DESCRIPTION:
We propose a trial to evaluate whether in-hospital glycemic control, as measured by mean daily glucose concentration and frequency of hypoglycemic events, is different between treatment with metformin and sitagliptin combination and treatment with glargine insulin once daily and rapid-acting insulin analog with meals in patients with type 2 diabetes. Hyperglycemia is associated with increased mortality, prolonged hospitalization and increased complications such as infection (1). Consensus guidelines recommend long-acting basal insulin and meal-time bolus insulin therapy for inpatient blood glucose management. These basal bolus regimens are labor intensive, require multiple injections each day, and can cause hypoglycemia. A study at our institution of patients admitted to the hospital and treated with our basal bolus insulin protocol found the incidence of hypoglycemia (blood glucose less than 70 mg/dl) to be 20% of all patient stays (2). A strategy for inpatient blood glucose management with less risk of hypoglycemia is needed.

We propose a trial of the use of two oral medications metformin and sitagliptin that lower blood sugar without the risk of hypoglycemia. Metformin is first-line therapy for outpatient management of type 2 diabetes. It has long-standing evidence of safety and efficacy. It decreases hepatic glucose production and increases insulin-mediated glucose utilization in the muscle and the liver. A Cochrane Review of 29 trials of metformin as monotherapy compared with other oral agents, insulin, diet, or placebo showed a reduction in cardiovascular events and all-cause mortality with metformin (3).

Sitagliptin is a Dipeptidyl-peptidase-4 (DPP-4) inhibitor approved by the FDA as monotherapy or in combination with metformin for the treatment of type 2 diabetes. Metformin and sitagliptin are active within 24 hours of initiation and do not cause hypoglycemia. Sitagliptin works by slowing the inactivation of glucagon-like peptide-1 (GLP-1). GLP-1 stimulates glucose dependent secretion of endogenous insulin with meals.

A recent preliminary study supports the use of sitagliptin for inpatient glucose management. This trial included 90 patients with type 2 diabetes admitted to general medicine and surgery services. It randomized patients to one of three groups: sitagliptin alone, sitagliptin plus long-acting insulin (glargine), or a basal bolus insulin regimen. The study selected for patients with mild to moderate diabetes by including only patients with diabetes controlled by diet alone, any combination of oral antidiabetic agents, or a total daily insulin dose ≤ 0.4 units/kg prior to admission. Patients were eligible if their blood sugar was 140 - 400 mg/dl. Patients in all three groups received supplemental (correction) doses of rapid-acting insulin before meals and bedtime for blood glucose >140 mg/dL. Glycemic control improved similarly in all treatment groups, but 100% of the patients in the sitagliptin alone group required one or more injections of rapid-acting insulin to correct hyperglycemia (4). This result suggests that sitagliptin alone is insufficient therapy for treating hyperglycemia in this population. We will recruit a similar population of patients, and we will add metformin for improved blood sugar control. Our sitagliptin and metformin group will not receive supplemental doses of rapid-acting insulin as the purpose of this trial is to evaluate a regimen without the risk of hypoglycemia.

Metformin is safe in patients with adequate renal function. The current prescribing information for metformin is that its use is permitted with a serum creatinine ≤ 1.4 mg/dL in women and ≤ 1.5 mg/dL in men which is equivalent to a GFR ≥ 60 ml/min (5). It is excreted by the kidneys and therefore can potentially accumulate in patients with renal failure. Metformin works by inhibiting gluconeogenesis-a process that utilizes lactic acid to produce glucose. Thus, with accumulation of this medication, it could predispose patients to lactic acidosis. The incidence of lactic acidosis with metformin is extremely low. A systematic review of 347 randomized trials and prospective cohort studies representing 70,490 patient-years of metformin use and 55,451 patient-years in the non-metformin group revealed no cases of lactic acidosis. Almost half of the studies allowed inclusion of patients with a serum creatinine above 1.5 mg/dL, and 97% of the studies allowed inclusion of patients with at least one contraindication to metformin therapy (6). Another trial evaluated the risk of lactic acidosis with metformin in 393 patients with renal insufficiency, with serum creatinine levels of 1.5 to 2.5 mg/dl (mean level 1.8 mg/dl) and found no cases of lactic acidosis over four years of the trial duration (7).

Most cases of lactic acidosis in patients taking metformin have been associated with shock or other tissue hypoxia. Elevated lactate in these patients may not be related to metformin. This is supported by the fact that lactic acidosis occurs as frequently in metformin users as users of other anti-diabetes medications (8). Also, metformin levels do not correlate with lactate levels or mortality suggesting that the underlying disease is more likely the cause of the acidosis than metformin (9). However this theoretical concern for an exceedingly rare complication has excluded metformin from use in hospitalized patients.

The recognition of the rarity of lactic acidosis among users of metformin with renal insufficiency has changed recommendations to allow for its use in patients with mild to moderate renal insufficiency. Current guidelines use an estimated GFR (eGFR) which is a more accurate approximation of renal function than serum creatinine. The current recommendation of the American Diabetes Association states that metformin can be used at full doses (2000 mg/day) as long as eGFR > 45 ml/min and serum creatinine is monitored. If the eGFR is < 45ml/min, then a maximal dose of 1000 mg/day is advised, with serum creatinine monitoring. Metformin should not be used if the eGFR is < 30 ml/min (10).

The American College of Radiology has recently updated their guidelines for the use of metformin in patients receiving IV contrast media (11). A prior guideline recommended holding metformin for 4 days surrounding IV contrast administration to evaluate for contrast-induced acute kidney injury. This guideline contributed to the practice of discontinuing metformin during hospitalization due to the commonness of radiology studies using IV contrast. There is no drug interaction between metformin and contrast media nor is there any effect of metformin on renal function. Given the risk of contrast-induced acute kidney injury is very low in patients with normal renal function and no co-morbidities, the revised (2013) American College of Radiology guidelines recommend that metformin can be continued without the need to evaluate renal function following contrast media. In the presence of co-morbidities that increase the risk for developing acidosis (liver dysfunction, alcohol abuse, heart failure, myocardial or peripheral muscle ischemia, sepsis or severe infection), the new guidelines recommend holding metformin for two days after IV contrast administration. Our study will only include patients without these co-morbidities and with normal renal function (eGFR > 60 ml/min). All subjects will have serum creatinine measured daily, and metformin will be discontinued in the event of acute kidney injury.

Since metformin is safe and effective for glucose management in patients with type 2 diabetes and normal renal function, we propose its continuation during hospitalization. This study will include adult patients with type 2 diabetes currently treated with metformin alone or in combination with other anti-diabetic agents including low dose insulin. All subjects will have normal renal function (eGFR>60 ml/min) and no comorbidities that increase the risk for acidosis. This prospective, randomized controlled trial will compare metformin and sitagliptin (which cannot cause hypoglycemia) to usual insulin therapy, which is known to cause hypoglycemia. This study has possible implications for improving the safety of therapy for hospitalized patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 80 years admitted to a general medicine services not requiring intensive care and not expected to require surgery.
2. Type 2 diabetes for ≥ 3 months treated with metformin (≥ 1000 mg/day) alone or metformin (≥ 1000 mg/day) with glimepiride, glyburide, glipizide, saxagliptin, sitagliptin, linagliptin, alogliptin, repaglinide, nateglinide, pioglitazone, exenatide, liraglutide, or a total daily dose of insulin ≤ 0.4 units/kg/day prior to admission.
3. Blood glucose>140 mg and < 400 mg/dL

Exclusion Criteria:

1. Acute critical illness expected to require admission to a critical care unit
2. Patients expected to require major surgery (requiring general anesthesia)
3. Patients expected to require gastrointestinal suction
4. Patients treated with less than 1000 mg/day of metformin prior to admission
5. Patients expected to be kept nothing by mouth (NPO) for >24-48 hours after admission
6. Patients with impaired renal function estimated GFR less than 60 ml/min based on the Modification of Diet in Renal Disease (MDRD) Study equation.
7. Clinically significant liver dysfunction or current alcohol abuse
8. Uncompensated heart failure
9. Myocardial or peripheral muscle ischemia
10. Sepsis or severe infection
11. Treatment with glucocorticoid greater than prednisone 5 mg daily or the equivalent
12. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
13. Pregnancy or breast-feeding at time of enrollment into the study

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
mean blood glucose for the duration of the hospital stay | duration of hospital stay
  Participants will be followed for the duration of the hospital stay, an expected average of 5 days.

SECONDARY OUTCOMES:
frequency of hypoglycemia | duration of hospital stay
  Participants will be followed for the duration of the hospital stay, an expected average of 5 days. The outcome is the percent of patients having any blood glucose value less than 70 mg/dl during their hospital stay.

OTHER OUTCOMES:
Acute kidney injury | duration of hospital stay
  Participants will be followed for the duration of the hospital stay, an expected average of 5 days. The outcome is the percent of patients who develop acute kidney injury during their hospital stay. Acute kidney injury is defined as an absolute increase in the serum creatinine concentration of ≥ 0.3 mg/dL from baseline or a percentage increase in the serum creatinine concentration of ≥ 50%